CLINICAL TRIAL: NCT03082482
Title: Smartphone-delivered Automated Video-assisted Smoking Treatment for People Living With HIV: Project AVAST - HIV
Brief Title: Smartphone-delivered Automated Video-assisted Smoking Treatment for People Living With HIV
Acronym: AVAST-HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7278
Record Dates: First submitted 2017-03-13; First posted 2017-03-17 (Actual); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Smoking Cessation
Keywords: Smoking Cessation; HIV; AIDS
MeSH Terms: conditions — Smoking Cessation; Acquired Immunodeficiency Syndrome | interventions — Tobacco Use Cessation Devices; Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Treatment (Active Comparator): Participants randomized to Standard Treatment will receive a smartphone with active service, brief advice to quit smoking (self-help materials), and 8-week supply of nicotine replacement therapy (patches), and provided 5 proactive phone counseling sessions by a trained Certified Tobacco Treatment Specialist.
  Interventions: Behavioral: Self-help materials; Drug: nicotine patch; Behavioral: Counseling
- Automated Treatment (Experimental): Participants randomized to Automated Treatment will receive smartphone-delivered automated treatment that will provide tailored smoking cessation treatment by way of video clips, text and graphical messages. Participants will receive notifications on the study provided smartphone once a week for an 8-week treatment period. Content delivered will be specific to the participants smoking status and motivation to quit.
  Interventions: Behavioral: Self-help materials; Drug: nicotine patch; Other: Smartphone-delivered automated treatment

INTERVENTIONS:
Behavioral: Self-help materials — Self-help smoking cessation materials
Drug: nicotine patch — Participants who smoke >10 cigarettes per day will receive 4 weeks of 21 mg, 2 weeks of 14 mg, and 2 weeks of 7 mg nicotine patches. Participants who smoke <10 cigarettes per day will receive 6 weeks of 14 mg and 2 weeks of 7 mg nicotine patches.
Behavioral: Counseling — Proactive phone counseling with a Certified Tobacco Treatment Counselor
  Arms: Standard Treatment
Other: Smartphone-delivered automated treatment — Tailored video clips, text and graphical messages delivered automatically each week to the participant.
  Arms: Automated Treatment

SUMMARY:
The proposed pilot study seeks to address the smoking treatment needs of people living with HIV/AIDS (PLWHA) by evaluating the feasibility and preliminary efficacy of a smartphone delivered automated video-assisted smoking treatment (AVAST). AVAST will enable smoking cessation treatment content to be presented with voice/audio, images, videos, and text in an interactive, structured format anytime and anywhere. This automated treatment approach is designed to enhance treatment engagement and facilitate abstinence from smoking among PLWHA. Participants will be recruited from the University of Oklahoma Health Sciences Center (OUHSC) clinics providing care to HIV+ individuals (e.g., the Infectious Diseases Institute).

DETAILED DESCRIPTION:
Substantial evidence indicates that the prevalence of cigarette smoking among persons living with HIV/AIDS (PLWHA) is far higher than the prevalence in the general US population. Moreover, strong associations between smoking and numerous adverse AIDS- and non-AIDS-related outcomes have been detailed. Thus, efficacious smoking cessation programs targeted to PLWHA are needed. Despite the need, relatively few smoking cessation intervention trials for PLWHA have been conducted, and the published results from these trials have not been overly positive. The currently available literature indicates that HIV+ smokers appear to be motivated to quit, as evidenced by high enrollment rates. Also, it appears that more intensive interventions result in significantly higher quit rates (vs. minimal interventions) at short term and intermediate follow-ups. However, smoking relapse rates are very high, and treatment effects are not well sustained. This study seeks to address this treatment need by evaluating the feasibility and preliminary efficacy of a smartphone-delivered automated video-assisted smoking treatment (AVAST).

Participants (n=20) will be randomized to one of two treatment conditions: 1) Standard Treatment (ST; n=10) or Automated Treatment (AT; n=10). In the ST condition, research staff will provide participants with in- person brief advice to quit and enroll them in a proactive telephone counseling program for smoking cessation. This ST approach mirrors the Ask Advise Connect (AAC) approach that our team has previously developed and implemented in numerous clinic settings. ST will be evaluated against AT, the fully automated AVAST approach. In the AT condition, smokers will be provided with in-person brief advice to quit and be enrolled in a fully automated and interactive smartphone-based treatment program that comprises interactive text messaging, images and audio/video clips. Participants in both treatment conditions will be provided with nicotine replacement therapy (NRT) in the form of transdermal patches. The goal of this pilot project is to establish the preliminary efficacy and feasibility of AT. Data collected in the pilot will then be used to support the submission of a NIH R01 application, and to determine if AT performs no worse than the more resource intensive ST approach. If lack of inferiority is established in the larger project, the AT approach will be readily scalable; easily implemented by community-based clinics and organizations; and offer an efficient way to allocate limited public health resources to tobacco control interventions.

ELIGIBILITY:
Inclusion Criteria:

* >/= 18 years
* Smoked >/= 100 cigarettes in a lifetime
* English speaking
* Currently smoking 5 or more cigarettes per day
* Willing to make a quit attempt within 1 week of enrollment
* HIV positive

Exclusion Criteria:

* History of medical condition that precludes the use of nicotine replacement therapy
* Current use of smoking cessation medications
* Pregnant or nursing
* Enrolled in another smoking cessation study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2017-05-19 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Smoking status by collecting an expired carbon monoxide breath sample | 3-Month Follow-Up
  Biochemically verifying smoking status on all participants by collecting an expired carbon monoxide breath sample.

SECONDARY OUTCOMES:
Participant satisfaction with treatment using the Client Satisfaction Questionnaire | 3-Month Follow-Up
  The investigators will use the Client Satisfaction Questionnaire to evaluate participant satisfaction.
Dropout rate | 3-Month Follow-Up
  The investigators will assess the number of participants who dropped out of the study.
Intervention delivery rate | 3-Month Follow-Up
  The investigators will assess the number of sessions completed by participants.

CONTACTS AND LOCATIONS:
Overall Officials: Damon Vidrine, DrPH, Principal Investigator — OUHSC
Locations (1):
- Oklahoma Tobacco Research Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Palmer MJ, Henschke N, Villanueva G, Maayan N, Bergman H, Glenton C, Lewin S, Fonhus MS, Tamrat T, Mehl GL, Free C. Targeted client communication via mobile devices for improving sexual and reproductive health. Cochrane Database Syst Rev. 2020 Jul 14;8(8):CD013680. doi: 10.1002/14651858.CD013680. PMID 32779730